CLINICAL TRIAL: NCT05242315
Title: Feasibility, Efficacy And Safety Of De Novo Extended-Release Tacrolimus Following Liver Transplantation
Brief Title: Extended-Release Tacrolimus Following Liver Transplantation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105029
Record Dates: First submitted 2022-01-19; First posted 2022-02-16 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Liver Transplant; Complications; Renal Insufficiency; Immunosuppressant Adverse Reaction; Metabolic Syndrome; Cardiovascular Diseases
MeSH Terms: conditions — Renal Insufficiency; Metabolic Syndrome; Cardiovascular Diseases | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Envarsus (Active Comparator): Envarsus tablet Dose 0.11 - 0.13 mg/Kg/day Frequency: once per day
  Interventions: Drug: Envarsus Oral Product
- Prograf (SOC) (Other): Prograf tablet Dose 0.10 - 0.15mg/Kg daily Frequency: 2 doses per day (dose above split in half for each dose)
  Interventions: Drug: Prograf (SOC)

INTERVENTIONS:
Drug: Envarsus Oral Product — as described in arm/group description
  Arms: Envarsus
Drug: Prograf (SOC) — Prograf (SOC)
  Arms: Prograf (SOC)

SUMMARY:
Medications used after transplant to prevent rejection are associated with many side effects. Tacrolimus side effects include kidney dysfunction; tremor, headaches, difficulty sleeping, change in sensation (legs), seizure, or confusion; high blood pressure; anemia, or low blood cell counts; diabetes; abnormal cholesterol and weight gain. The investigators want to use a new, approved, formulation of the standard medication (Envarsus) as they believe it may be associated with reduced side effects. The investigators would like to assess how safe it is to use this medication and how well it works in comparison to currently used formulations. The investigators will study if there are less side effects and will study clinical outcomes (including how well the liver does and if there is need for hospitalizations after transplant).

The investigators hope that this information will improve the care provided to and outcomes in patients following liver transplant.

DETAILED DESCRIPTION:
PURPOSE

To assess the impact of Envarsus on toxicity and clinical outcomes in participants following liver transplant. Tacrolimus-based immunosuppression is the standard of care following liver transplantation (LT). This medication is associated with significant toxicity including renal dysfunction, increased risk of diabetes and neurotoxicity. Of note, both nephrotoxicity and neurotoxicity occur at elevated peak serum tacrolimus blood concentrations and improve when the dose is reduced or discontinued. Envarsus does not have the high peak seen with initial dosing in the other formulations. This may be one of the reasons Envarsus use improves tremor associated with tacrolimus use.

HYPOTHESES

Use of extended-release tacrolimus following LT will be: 1. Effective and safe. 2. Without any difference in rejection. 3. Less nephrotoxic with reduced incidence of renal impairment. 4. Better with regard to features of metabolic syndrome including myosteatosis. 5. Less neurotoxic. 6. Better with regard to both graft and patient survival when compared to immediate-release tacrolimus (Prograf®).

JUSTIFICATION

Tacrolimus-associated toxicity, especially renal dysfunction is common following LT (up to 25%) and is associated with increased mortality. Showing extended-release tacrolimus (Envarsus) is safe and efficacious will lead to broader use in the post-transplant setting. Use of this regimen leads to decreased maximum concentration and in some studies has shown benefit with regards to renal function. Such benefit will no doubt translate into improved long-term outcomes including survival and reduced healthcare costs.

OBJECTIVES/AIMS

The aim of this study is to assess the feasibility, safety and efficacy of using Envarsus in comparison to the immediate-release tacrolimus (Prograf®) following LT. Additional objectives include impact on renal function, metabolic syndrome, myosteatosis (fatty infiltration of skeletal muscle; reflects poor quality and function and correlated with poor outcomes), cardiovascular events, neurotoxicity, graft and patient survival.

METHODS

Basic study design

This will be a randomized control trial where participants will be randomized 1:1 to two groups: i) Prograf (dose 0.10 - 0.15mg/Kg daily; divided into BID dosing), ii) Envarsus (0.11 - 0.13 mg/Kg/day); both groups will be on mycophenolate (dose 1g BID) and will receive basiliximab (dose 20 mg) for induction at POD 0 and 4. Participants will be enrolled prior to transplant or up to 90 days following LT. The first dose will be administered within 90 days of LT. Randomization will be done at the first post-transplant outpatient visit (30-90 days post-transplant). Randomization will be stratified according to gender, bilirubin (< 50 and ≥ 50 umol/L), albumin (<30 and ≥ 30 g/L) and diagnosis of diabetes and renal function (according to the category of estimated GFR (45 to <60 ml, or 60 to <90 ml per minute per 1.73 m2)) to ensure that all groups are homogeneous. Tacrolimus will be taken orally with water, twice daily in the immediate-release group and once daily in the extended-release group for the duration of the study. Participants will take tacrolimus at approximately the same time each day (1 hour before meals). Participants will be instructed to swallow the tablet whole (no chewing, dividing, or crushing the tablet).

All participants who have received a liver transplant at the University of Alberta in Edmonton, Canada who are at least 18 years of age will be eligible for enrollment (18 month period following study initiation).

The primary analysis will be at 1-year, however, there will be a 10 year period of follow up off-trial. This will include participant outcomes (hospitalizations, complications of rejection, diabetes, renal dysfunction, cardiovascular events, graft and participant survival). The study will be carried out in compliance with the International Conference on Harmonization Harmonized Tripartite Guideline for Good Clinical Practice.

Covariates of interest

Baseline participant characteristics - Participant demographics; height, weight, BMI and waist circumference; etiology of cirrhosis; co-morbidities including diabetes, dyslipidemia, hypertension, smoking status and cardiovascular disease. History of malignancies at the time of transplant evaluation will also be noted. Immunosuppression (IS) following LT (at discharge, 1-, 3-, 6-, 12-, 60-months following LT and at end of follow up) and levels and dose of IS will also be recorded. Any changes, or adverse events including neurotoxicity due to IS will also be recorded. Finally, any episodes of rejection (based on biopsy) will be recorded. Biopsy will be obtained if clinically indicated at any time during the post-transplant course based on the participants presentation (persistently elevated liver enzymes or liver function tests, or abnormal FibroScan (liver stiffness > 9 kPa)). FibroScan will be done at one year, two years post-transplant and then every 2-years until end of follow up.

Biochemistry - serum creatinine, INR, sodium and bilirubin will be acquired. Data on albumin, transaminases, GGT, electrolytes, and CBC will also be collected. Values for lipid profiles, random and fasting blood glucose, insulin levels, and hemoglobin A1C will be recorded.

Analysis plan

Safety and efficacy - will be assessed descriptively. All participants who received at least one dose of Envarsus® will be included for analysis in the Envarsus® group. Only treatment related adverse events will be analyzed (complications following surgery such as bile leak, vascular thrombus, etc. will not be reported). The difference between the groups with regards to number of adverse events will be determined using poisson regression.

Incidence of acute rejection will be reported; Cox regression will be used to determine if there is a difference between the 2 study groups.

Impact of extended-release tacrolimus on secondary endpoints:

Impact on renal function - Proportion of participants with renal impairment (change in GFR 10%), number of episodes of AKI, incidence of AKI and CKD will be reported. The investigators will use Cox regression to determine if there is a difference between the 2 study groups with regards to renal function. Participants will be analyzed according to the treatment group to which they were randomized and not based on medication taken during the course of the study.

Incidence of diabetes, metabolic syndrome, and neurotoxicity will be reported. Rates of hospitalization, incidence of myosteatosis and patient and graft survival will be reported. Cox regression will be used to determine if there is a difference between the 2 study groups with regards to neurotoxicity and development of myosteatosis. The investigators will use poisson regression to determine difference between groups with regards to hospitalization rates. The investigators will use ANCOVA to determine if there is a difference between groups with regards to features of metabolic syndrome (diabetes, glycemic control, dyslipidemia, weight gain and hypertension). Difference in LOS between groups will be determined using linear regression. The investigators will use Kaplan Meier curves and log-rank test to determine if there is a difference in graft survival or mortality between the two arms (p-value will be provided).

Sample size calculation

This is a feasibility study thus no sample size calculation was required. The investigators will aim to enroll 94 participants over a 18 month period. Recruitment should not be a problem as approximately 90-100 LT are done each year at the University of Alberta.

ELIGIBILITY:
Inclusion Criteria:

- Adult individuals transplanted at the University of Alberta

Exclusion Criteria:

* Individuals with congenital long QT syndrome
* Patients with elevated bilirubin > 100 umol/L post-LT (at day 3)
* Patients with chronic kidney disease (eGFR < 45 ml per minute per 1.73 m2)
* Patients with acute kidney injury requiring discontinuation of calcineurin inhibitors.
* Patients who have hepatocellular carcinoma, require a re-transplant, or receive multi-visceral transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2034-02-15 (Estimated)

PRIMARY OUTCOMES:
Safety of Envarsus as indicated by adverse events | 1 year
  Adverse events include frequency of transplant rejection, and changes from baseline in clinical laboratory parameters

SECONDARY OUTCOMES:
Incidence of renal impairment | 1-10 years
  We will consider participants with >10% decline in GFR to represent a group with renal impairment. We will define acute kidney injury (AKI) as at least a 50% and/or a 26.5 µmol/L (0.3 mg/dL) increase in serum creatinine level relative to the baseline reference value as per Kidney Disease: Improving Global Outcomes (KDIGO) criteria (11) in participants without pre-existing CKD. CKD will be defined as eGFR <60 ml/min for more than 3 months, according to the KDIGO criteria (13), evidence of intrinsic renal disease or requiring renal replacement therapy. Acute on CKD will be defined as at least a 50% and/or a 26.5 µmol/L (0.3 mg/dL) increase in serum creatinine level relative to the baseline reference value as per KDIGO criteria (11) in participants with pre-existing CKD. The baseline creatinine will be defined as the minimum of all values available within 3 months of LT.
Number of patients with metabolic syndromes [diabetes] | 1-10 years
  Diabetes will be diagnosed based on an elevated fasting plasma glucose (≥7.0 mmol/l) or an elevated 2-hour plasma glucose (≥11.1 mmol/l) during an oral glucose tolerance test or an elevated random plasma glucose (≥11.1 mmol/l).
  Glycemic control will be measured by fasting blood glucose and hemoglobin A1C (at 3-, 6-, 12, 60-months following LT and at end of follow up). Change in hemoglobin A1C at 1 year post LT from baseline will be used as a measure of glycemic control. Hemoglobin A1C value within 3 months of LT will be used as the baseline value.
Incidence of neurotoxicity | 1 years
  adverse events including tremor, headache, insomnia, dysesthesia, or mood disturbance will be recorded. Severe events including akinetic mutism, seizures, cortical blindness, focal neurological deficits, encephalopathy, decreased cognitive ability and psychosis will be monitored and recorded
Length of stay in hospitalized patients | 1-10 years
  From time of admission for surgery to time of discharge.
Incidence of Intensive Care Unit (ICU) admission | 1-10 years
  Looking at if the patient is admitted to the ICU post transplant
Length of Intensive Care Unit admission | 1-10 years
  Length of stay in the intensive care unit if admitted post transplant
Incidence of hospitalizations | 1-10 years
  how many patients are hospitalized post transplant
Patient Survival | 1-10 years
  Liver-related versus all-cause mortality will be documented.
Graft Survival | 1-10 years
  Any re-transplants will be recorded.
Impact on quality of life (QOL) - Chronic Liver Disease Questionnaire | 1 year
  Using the Chronic Liver Disease Questionnaire (CLDQ) which is a disease specific questionnaire. This will be administered twice during the study period; at the start and after 12 months of study enrollment.
  Minimum score: 1 Maximum score: 7
  The higher score indicates a better outcome
Impact on quality of life (QOL) - EuroQuol-5Dimensions-5 Levels Questionnaire | 1 year
  EuroQuol-5Dimensions-5Levels (EQ-5D-5L)
  Description System section Maximum score 1 Minimum score 5
  A higher score indicates a lower assessment for quality of life
Muscularity assessment | 1 year
  mean muscle attenuation in Hounsfield units will be calculated for the entire muscle area at the third lumbar (L3) vertebra. Myosteatosis will be defined as <41 mean Hounsfield units in patients with a BMI up to 24.9, and <33 mean Hounsfield units in those with a BMI ≥25. These cut-off values have been used previously in patients with cirrhosis and have been shown to be associated with mortality (17). We will use CT L3 skeletal muscle index (L3 SMI) expressed as cross sectional muscle area/height2, and cutoffs for sarcopenia will be based on values for cirrhotic patients (L3 SMI: < 39 cm2/m2 for women and < 50 cm2/m2 for men). CT will be obtained at 1 year post-LT.
Impact on quality of life (QOL) - EuroQuol Visual Analogue Scale (VAS) | 1 year
  EuroQuol Visual Analogue Scale (VAS) Max score 100 Minimum score 0
  A higher score indicates a higher quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Univerity of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Potential to share de-identified data if requested from other researchers.